CLINICAL TRIAL: NCT05249413
Title: Outcomes of Early Vitrectomy for Endophthalmitis After Cataract Surgery in Delta Population, Egypt, 2015-2020.
Brief Title: Early Vitrectomy for Endophthalmitis After Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Other Study IDs: RC-14-2-02
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Endophthalmitis; Cataract; Vitreous Detachment; Retinal Detachment
Keywords: endophthalmitis; cataract; vitrectomy; retinal detachment
MeSH Terms: conditions — Endophthalmitis; Cataract; Vitreous Detachment; Retinal Detachment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endophthalmitis after primary cataract surgery.: Cases diagnosed as acute post-operative endophthalmitis after primary cataract surgery.
  Interventions: Procedure: Early 23-gauge pars-plana vitrectomy

INTERVENTIONS:
Procedure: Early 23-gauge pars-plana vitrectomy — pars-plana vitrectomy for management of acute post-operative endophthalmitis.

SUMMARY:
Post-operative infectious endophthalmitis is devastating condition that causes a diffuse intraocular inflammation and may lead to blindness. Acute post-operative endophthalmitis usually presented within 6 weeks of intraocular procedure and diagnosis is confirmed by clinical examination and by the aid of B-scan ultrasonography.

DETAILED DESCRIPTION:
There is no consensus regarding the timing of vitrectomy in cases with endophthalmitis after cataract surgery. The Endophthalmitis Vitrectomy Study concluded that vitrectomy should be preserved for cases with only light perception. The advances in posterior segment machines and small gauge cannulas decrease the incidence of intra-operative complications and encourage for early intervention in cases with endophthalmitis after primary cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset endophthalmitis within 6 weeks after primary cataract surgeries.
* Patients had undergone early pars-plana vitrectomy within 48 hours of their confirmed diagnosis.

Exclusion Criteria:

* Patients were diagnosed as endogenous or chronic endophthalmitis.
* Patients with a previous history of rupture globe surgery or trauma.
* Patients who didn't complete the follow up period.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that were diagnosed as acute post-operative endophthalmitis at ophthalmology department, Benha University Hospital, EGYPT.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity | Baseline and 3 months after intervention.
  Changes in visual acuity from baseline and after early vitrectomy operation.

SECONDARY OUTCOMES:
Other prognostic factors | Baseline and 3 months after intervention.
  Other factors that may influence the final visual outcome in cases with endophthalmitis as (intraocular tamponade, posterior vitreous detachment, systemic condition and virulence of causative organism)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdelshafy, MD, Study Chair — Benha University
Locations (1):
- Ophthalmology department, Benha University, EGYPT, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Undecided